CLINICAL TRIAL: NCT06042114
Title: The Effect of Listening to Surah Al-Inshirah on Pain and Anxiety After Laparoscopic Cholecystectomy Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seher Tanrıverdi (Other)
Responsible Party: Sponsor-Investigator, Seher Tanrıverdi, Asistant Professor, Mardin Artuklu University
Organization: Mardin Artuklu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mardin-Artuklu University
Record Dates: First submitted 2023-09-08; First posted 2023-09-18 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Patients of Laparoscopic Cholecystectomy
Keywords: Laparoscopic Cholecystectomy; postoperative; pain; Surah Inshirah; anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Listening to Surah Inshirah (Experimental): Experimental group patients; A patient descriptive characteristics form will be applied, pretest VAS pain score and state anxiety scale will be applied. Then, the Surah al-Inshirah will be listened to and the final test VAS pain score and state anxiety scale will be applied.
  Interventions: Behavioral: Surah Inshirah
- control group (No Intervention): Control group patients; A patient descriptive characteristics form will be applied, pretest VAS pain score and state anxiety scale will be applied. The posttest VAS pain score and state anxiety scale will be applied 10 minutes later, without any intervention.

INTERVENTIONS:
Behavioral: Surah Inshirah — Patients in the experimental group will be listened to the Surah al-Inshirah after surgery and its effect on pain and anxiety levels will be evaluated.
  Arms: Listening to Surah Inshirah

SUMMARY:
In the postoperative period, good pain and anxiety management is required to minimize complications and ensure recovery. Patients should be evaluated with a holistic approach, taking into account factors such as physical and psychological discomfort, anxiety level, age, gender, previous pain level. Pharmacological and non-pharmacological methods are used to relieve pain and anxiety in the postoperative period.

Non-pharmacological methods reduce the patient's pain and anxiety by creating a feeling of comfort and control in the patient. Relaxation techniques such as hypnosis, yoga and music are among these. The main purpose of these methods is to draw the attention of the individual in another direction. Praying is also one of the non-drug methods, and the number of studies on this subject is very limited, and there are studies where it has been determined that praying and praying reduces the anxiety levels of patients.

Purpose To examine the effect of listening to Surah al-Inshirah on pain and anxiety after laparoscopic cholecystectomy surgery.

Method The population of the study will consist of patients who have undergone laparoscopic cholecystectomy at Mardin Training and Research Hospital and Kızıltepe State Hospital, who meet the inclusion criteria and volunteer to participate in the research.

The study group of 60 people who will participate in the research will be divided into two equal groups according to the table of random numbers obtained from the computer-based Research Randomizer program.

Experimental group patients; A patient descriptive characteristics form will be applied, pretest VAS pain score and state anxiety scale will be applied. Then, the Surah al-Inshirah will be listened to and the final test VAS pain score and state anxiety scale will be applied.

Control group patients; A patient descriptive characteristics form will be applied, pretest VAS pain score and state anxiety scale will be applied. The posttest VAS pain score and state anxiety scale will be applied 10 minutes later, without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can be contacted,

  * Patients with an abdominal pain score of 4 and above as evaluated by VAS after laparoscopic cholecystectomy surgery,
  * Patients aged 18 and over were included in the study.

Exclusion Criteria:

* Patients who can be contacted,

  * Patients with an abdominal pain score of 4 and above as evaluated by VAS after laparoscopic cholecystectomy surgery,
  * Patients aged 18 and over were included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2023-10-19 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Patient Information Form | It will be applied to patients in the clinic 2 hours before the laparoscopic cholecystectomy procedure
  This form, created by the researcher with the support of the relevant literature, consists of 9 questions that question the patients' education level, age, gender, occupation, marital status, income level, previous surgery experience and coping methods used for pain and anxiety in daily life.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from initial Visual Analog Scale in 10 minutes
  The patient was asked to mark on a 10 cm horizontal line showing his current status on the Visual analog scale. In this study, for pain and anxiety; Markings were made on a 10 cm horizontal line, one end indicating that the patient's pain was very good (0 = no pain), and the other end indicating that the patient's pain was very bad (10 = most severe). The distance from the point where there was no pain or anxiety (0) to the point marked by the patient was measured. The value found shows the patient's pain and anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: SEHET TANRIVERDİ, PhD, Principal Investigator — Mardin Artuklu University
Locations (1):
- Mardin State Hospital, Mardin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
can be reviewed by other researchers after the study has been published.

REFERENCES:
- [Background] Naimi E, Eilami O, Babuei A, Rezaei K, Moslemirad M. The Effect of Religious Intervention Using Prayer for Quality of Life and Psychological Status of Patients with Permanent Pacemaker. J Relig Health. 2020 Apr;59(2):920-927. doi: 10.1007/s10943-018-0698-8. PMID 30218372
- [Result] Acar, K., Aygin, D. (2016). Laparoskopik cerrahi sonrası ağrı ve hemşirelik bakımı. Online Türk Sağlık Bilimleri Dergisi, 1(2), 17-22.
- [Result] Çakır, H.S.K., Yılmaz, Ü.D. (2018). Laparoskopik kolesistektomi uygulanan hastaların taburculuk öncesi bilgi gereksinimlerinin belirlenmesi. Türkiye Klinikleri Dergisi, 10(2), 115-121.
- [Result] Cimilli, C. (2001). Cerrahide anksiyete. Klinik Psikiyatri, 4(3), 182-186. Erişim 27.08.2019, https://www.journalagent.com/kpd/pdfs/KPD_4_3_182_186.pdf